CLINICAL TRIAL: NCT03283943
Title: Phase I (Safety Assessment) of Durvalumab (MEDI4736) With Focal Sensitizing Radiotherapy in Platinum Resistant Ovarian, Primary Peritoneal or Fallopian Tube Epithelial Carcinoma
Brief Title: PDL-1 Inhibition and Focal Sensitizing Radiotherapy in Recurrent Ovarian/Primary Peritoneal/Fallopian Tube Cancers.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Ozmosis Research Inc. (Industry)
Responsible Party: Principal Investigator, Anna Tinker, Medical Oncologist, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-078
Record Dates: First submitted 2017-06-30; First posted 2017-09-15 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab and focal radiotherapy (Experimental): Durvalumab 1500 mg IV every 28 days, and 2 fractions of focal sensitizing radiation with cycles 1 and 2 of treatment.
  Interventions: Radiation: Focal radiotherapy; Drug: Durvalumab

INTERVENTIONS:
Radiation: Focal radiotherapy — Focal sensitizing radiotherapy will be given at a starting dose level of 24 Gray (6 Gy X 4 fractions), and may be escalated to 32 Gy (8Gy X4 fractions).
Drug: Durvalumab — Durvalumab 1500 mg IV every 28 days
  Other Names: MEDI 4736

SUMMARY:
It is postulated that focal sensitizing radiotherapy may potentiate the effectiveness of durvalumab. The purpose of this study is to test the safety and tolerability of 2 different dose levels of focal sensitizing radiation therapy given with durvalumab.

DETAILED DESCRIPTION:
Durvalumab is a PDL-1 inhibitor, part of class of agents (called checkpoint inhibitors) designed to increase the ability of the immune system to recognize and work to eliminate cancers. Checkpoint inhibitors have been studied in recurrent ovarian, primary peritoneal and Fallopian cancers, and on their own show a low level of activity.

Radiation therapy is usually used in women with recurrent ovarian, primary peritoneal and Fallopian cancers to palliate symptoms related to progressive disease. However, radiation is know to modify the cancer immune environment and to release tumour antigens. These actions may potentiate the function of immune checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study specific procedures
* Female patients aged 19 years and older
* Platinum-resistant (progression within 6 months of platinum based regimen) or platinum-refractory ovarian/fallopian tube/peritoneal origin.
* High grade serous, endometrioid, clear cell, mucinous, malignant mixed Mullerian tumor, and low grade serous histotypes are permitted. Non-epithelial tumours will not be permitted.
* ECOG performance status 0-1.
* No more than 2 lines of therapy in the platinum-resistant setting.
* No bowel obstructions within the preceding 6 months.
* Last radiation therapy treatment ≥3 months prior to enrollment.
* Expected survival >3 months.
* All patients much have at least one site of measurable disease as defined by RECIST criteria (v.1.1).
* All patients must have disease suitable for core biopsy and agree to study related biopsies. Disease suitable for biopsy can serve as radiation targets, but cannot be used for response assessment.
* All patients must have at least 2 additional sites of disease that serve are suitable radiation targets (see section 6.2.1).
* Lesions suitable for radiation targeting must meet all of the following criteria:
* each target must be > 4 cc in volume by standard imaging techniques, such as CT scan, MRI, or radiograph
* for each lesion, partial treatment of a tumour mass is permitted, but the treatment volume cannot be less than the equivalent of a 2cm sphere (4cc) and the two targets cannot be part of the same contiguous mass
* must be outside of previously irradiated fields 12. Adequate organ and marrow function

Exclusion Criteria:

* Subjects who cannot meet all the radiation planning constraints will not be eligible for this trial.
* Participation in another clinical study with an investigational agent during the last 4 weeks.
* Concurrent enrolment in another clinical study, the only exception being observational (non-interventional) clinical studies.
* History of pneumonitis requiring treatment with steroids, or has a history of interstitial lung disease.
* Patients who have contraindications to receiving radiation therapy, such as: Rheumatoid Arthritis, connective tissue disorders, Lupus, scleroderma, CREST syndrome, Crohn's syndrome, Ulcerative colitis, or other conditions identified by the Radiation Oncologist as unsuitable for radiation therapy.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of the study drug, with the exception of intra-nasal and inhaled corticosteroids or systemic corticosteroids at physiologic doses, which must not exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Prior exposure to an anti-PD-1 or anti-PD-L1 antibody.(including durvalumab
* History of acute diverticulitis, intra-abdominal abscess, or GI obstruction.
* Previous severe hypersensitivity reaction to another monoclonal antibody (mAb).
* Active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with Vitiligo, Grave's disease or psoriasis not requiring systemic treatment (within the past 2 years) or those with resolved childhood asthma/atopy are not excluded.
* Uncontrolled intercurrent illness including: infection requiring therapy, symptomatic congestive heart failure, uncontrolled hypertension (systolic blood pressure > 150 and diastolic blood pressure >100), unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses.
* Mean QT interval corrected for heart rate (QTc) ≥ 470 ms calculated from using Frediricia'sCorrection.
* Positive for Human Immunodeficiency Virus (HIV), Hepatitis B (Hepatitis B Surface Antigen [HBsAg] reactive), or Hepatitis C virus (Hepatitis C Virus Ribonucleic Acid [HCV RNA] (qualitative) is detected).
* Previous clinical diagnosis of active tuberculosis.
* Receipt of a live attenuated vaccination within 30 days of study entry or within 30 days or receiving the study drug.
* History of another malignancy, with the exception of:
* Malignancy treated with curative intent without evidence of recurrence for ≥ 5 years
* Adequately treated non -melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease e.g. cervical carcinoma in situ
* Female patients who are pregnant, breast-feeding or of childbearing potential who are not employing an effective method of birth control (see Table 3).
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the study drug or interpretation of patient safety or study.

Ages: 19 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-12-16 (Estimated); Study Completion 2020-12-16 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of durvalumab combined with focal irradiation for use in recurrent ovarian cancer | First 4 weeks of therapy
  The maximum tolerated dose will be defined by dose-limiting toxicities and serious adverse events.

SECONDARY OUTCOMES:
Objective response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Objective Response rate as evaluated by RECIST (v 1.1) criteria 2) Progression free survival 3) Overall survival
CA-125 response rate | From date of study enrollment until confirmed CA-125 progression, through study completion, an average of 1 year
  Using GCIG CA-125 response criteria
Immune-related response rate | From date of study enrollment until confirmed immune-related disease progression, through study completion, an average of one1year
  Using Immune-related response criteria

OTHER OUTCOMES:
Survival | From date of study enrollment until death or study completion (maximum 12 months).
  Progression free survival and overall survival of the study population

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT03283943/Prot_000.pdf